CLINICAL TRIAL: NCT02621242
Title: Effects of the Anti-HIV Pill Truvada on Gene Transcription in the Gastrointestinal Tract of HIV-uninfected Individuals
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Joanne Stekler, MD MPH, Associate Professor, Division of Allergy & Infectious Diseases, University of Washington
Other Study IDs: 49167
Record Dates: First submitted 2015-11-10; First posted 2015-12-03 (Estimated); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-01

CONDITIONS: HIV
MeSH Terms: interventions — Gastroscopy; Proctoscopy; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: All subjects will undergo all procedures
  Interventions: Procedure: Upper endoscopy; Procedure: Anoscopy; Drug: Truvada

INTERVENTIONS:
Procedure: Upper endoscopy — Upper endoscopy with biopsies
Procedure: Anoscopy — Anoscopy with biopsies
Drug: Truvada — Truvada (tenofovir/emtricitabine) daily as HIV pre-exposure prophylaxis. This medication will not be provided by the study.

SUMMARY:
As explained in detail in a recently published hypothesis article (Hladik F. A new hypothesis on HIV cure. F1000Research, 4:77 (2015)), the investigators hypothesize that NRTI drugs may reduce the likelihood of HIV eradication by promoting the survival of cells with integrated provirus. In this study, the investigators will test whether daily oral use of two NTRI drugs, tenofovir and emtricitabine (Truvada Pill), induces changes in the upper and lower gut mucosa that are congruent with supporting this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* • HIV-negative

  * Male gender at birth
  * Age ≥18 years old
  * Intent to initiate PrEP in the next 1-2 months.
  * Willingness and ability to provide informed consent for study participation
  * Willingness to undergo all required study procedures

Exclusion Criteria:

* Creatinine clearance < 60mL/min
* Platelet count below the normal reference
* Coagulation (PT/PTT) tests above the normal reference
* Any prior use of PrEP
* Use of PEP within 30 days prior to study entry
* Receipt of

  * anti-coagulant medications (e.g. warfarin). Aspirin is allowable.
  * Systemic corticosteroid medications
  * Non-steroidal anti-inflammatory drug (NSAID) use >2 days/week
* Signs or symptoms of acute HIV infection within 14 days of study entry
* No availability of another person who will drive participant home on days of entry and follow-up procedures.
* Plan to leave the Seattle area in the subsequent 2.5 months
* Any condition or substance use that, in the opinion of the study investigator, would interfere with study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is a prospective observational study of cis-gender male persons initiating HIV pre-exposure prophylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Stekler, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort
Started | 9
Completed | 8
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cohort
Number analyzed (Participants) | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [28 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Global Transcriptome Analysis
Description: Global transcriptome analysis tests for expression changes of any possible gene across the entire human genome in response to Truvada PrEP. The main outcome of such an analysis is the number of genes significantly changing in expression between before and after treatment. We will report that Truvada PrEP up-regulates X number of genes and down-regulates Y number of genes.
Time Frame: 2-3 months after initiating HIV Pre-exposure prophylaxis
Population: Duodenal biopsies
Measure: Number; unit: genes
Units Other Than Participants: Genes
Arm/Group | Cohort
Number analyzed (Participants) | 8
Number analyzed (Genes) | 16321
genes
  Up-regulated | 116
  Down-regulated | 135

ADVERSE EVENTS:
Time Frame: Duration of study enrollment, approximately 2 months
Description: Serious adverse events would have been collected as part of the protocol, however, given that this was not an intervention study, only adverse events that might have been attributed to study procedures (i.e. specimen collection) would have been reported, had any occurred.
Arm/Group | Cohort
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT02621242/Prot_SAP_001.pdf